CLINICAL TRIAL: NCT04015674
Title: Effects of Aerobic Exercise on the Vascular Caliber of the Arteriovenous Fistula in Patients With Chronic Kidney Disease on Hemodialysis: a Randomized Cross-over Study
Brief Title: Effects of Aerobic Exercise on Arteriovenous Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 02867318.9.0000.5327
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Chronic Kidney Diseases
Keywords: Exercise; Vasodilation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Aneurysm | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Patients will remain in supine position for 5 minutes to measure their vascular caliber of the AVF by echography. After, will be instructed to perform 30 minutes on stationary bicycle (Model Monark). The AVF vascular caliber will be measured during aerobic exercise. Because it is a cross-over trial, participants will perform the other arm after 7 days.
  Interventions: Other: Exercise group; Other: Control group
- Control group (Active Comparator): The patients will perform 30 minutes of rest in a chair and the measurements will be performed in the same moments established by the exercise group. Because it is a cross-over trial, participants will perform the other arm after 7 days.
  Interventions: Other: Exercise group; Other: Control group

INTERVENTIONS:
Other: Exercise group — Aerobic exercise on a stationary bicycle
Other: Control group — In a rest

SUMMARY:
Arteriovenous fistula (AVF) is considered the gold standard for safe and effective vascular access during hemodialytic treatment. It is known that systemic aerobic exercise is capable of promoting peripheral vasodilation, however, its effects on AVF are unknown. For this reason, we will evaluate the effects of aerobic exercise on a stationary bicycle over the AVF caliber.

DETAILED DESCRIPTION:
Hemodialysis is a method responsible for filtering blood and helping to control excess blood fluid and impurities in patients with end-stage chronic kidney disease. The vascular accesses commonly used in this procedure is atribute catheter, which is placed in a large caliber vein, usually jugular or femoral vein, and arteriovenous fistula (AVF). In order to use the AVF in the hemodialysis procedure, a maturation process of the AVF is necessary, characterized by the increase of its caliber, which is accelerated by force exercises located in the AVF region, whose purpose is to promote the vasodilation of the AVF. Systemically performed aerobic exercises are also capable of promoting peripheral vasodilation and their effects on AVF are still unknown. Therefore, this study proposes to evaluate the behavior of the AVF through ultrasound before, during and after performing aerobic exercise on a stationary bicycle. For this, all patient will sign the informed consent form, respond to the International Physical Activity Questionnaire (IPAQ) and questionnaire Kidney Disease Quality of Life (KDQOL-SFTM), and use a pedometer for 7 days to measure the number of steps per day to characterize the sample. Patients will remain in supine position for 5 minutes to measure their vascular caliber of the AVF by echography. After, will be instructed to perform 30 minutes on stationary bike (Model Monark). The AVF vascular caliber will be measured during aerobic exercise. Because it is a cross-over trial, participants will perform the other arm after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who use AVF hemodialysis for at least 1 month.
* Patients on hemodialysis 3 times a week at the HCPA Nephrology Service.
* Age equal to or greater than 18 years.
* Physical conditions to perform exercises proposed in this study.
* Stability of chronic kidney disease for at least 30 days, defined by absence of hospitalization.

Exclusion Criteria:

* Acute myocardial infarction in the last 3 months.
* Acute infectious or inflammatory process.
* Decompensated coronary artery disease.
* Symptomatic peripheral arterial disease.
* Arteriovenous fistula in lower limbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-01-02 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Arteriovenous fistula caliber | 30 minutes
  The arteriovenous fistula caliber will be measured using ultrasound.

SECONDARY OUTCOMES:
Arterial pressure of carbon dioxide (PaCO2) | after 30 minutes of exercise or rest
  Gasometry
Arterial oxygen pressure (PaO2) | after 30 minutes of exercise or rest
  Gasometry

OTHER OUTCOMES:
Creatinine | after 30 minutes of exercise or rest
  Serum levels
Urea | after 30 minutes of exercise or rest
  Serum levels
phosphorus | after 30 minutes of exercise or rest
  Serum levels
potassium | after 30 minutes of exercise or rest
  Serum levels
sodium | after 30 minutes of exercise or rest
  Serum levels
calcium | after 30 minutes of exercise or rest
  Serum levels
blood count | after 30 minutes of exercise or rest
  Serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rovedder, PhD, Study Director — UNIVERSIDADE FEDERAL DO RIO GRANDE DO SUL (UFRGS)
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grade Do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No